CLINICAL TRIAL: NCT02112201
Title: Preventing HIV/STI Risk Behavior in Girls With Delinquency, Drug Abuse, & Trauma
Brief Title: The ProGirls Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DA025857
Record Dates: First submitted 2014-04-03; First posted 2014-04-11 (Estimated); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Delinquency; HIV Risk; Substance Use; Trauma Exposure
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Integrated intervention for parents and adolescent girls (Experimental): Twelve session parent education and support group; twelve session one-on-one adolescent skills training intervention
  Interventions: Behavioral: Integrated intervention for parents and adolescent girls
- Treatment as usual (No Intervention): Treatment as usual

INTERVENTIONS:
Behavioral: Integrated intervention for parents and adolescent girls — The intervention will consist of individually administered preventive curriculum for adolescent girls involved in the juvenile justice system that integrally addresses delinquency, drug abuse, and trauma exposure, along with group-based training and support for parents.
  Arms: Integrated intervention for parents and adolescent girls

SUMMARY:
Girls in the juvenile justice system who have high rates of delinquency, drug abuse, and trauma are particularly at risk for engaging in risky sexual behavior and for contracting HIV/AIDS or other sexually transmitted infections (STIs). No effective prevention programs for girls who have this combination of behaviors is known to exist at this time. Researchers are developing, assessing, and implementing a family-centered prevention program to decrease girls' participation in the risky behaviors associated with the spread of HIV and STIs. The program also includes a group-based training and support program for parents.

DETAILED DESCRIPTION:
This study aims to test an intervention to reduce HIV/STI risk behavior among girls in the juvenile justice system with the triple-threat risk of delinquency, drug abuse, and trauma. This is a competing continuation of the ProTeens study (Preventing Drug Abuse & HIV/AIDS in Delinquent Youths: An Integrated Intervention) which focused on testing a family-centered intervention for treating HIV risk, drug use, and delinquency in boys. The current study will adapt the ProTeens intervention for girls. Girls and their parent(s) will be randomly assigned to either a family-centered intervention condition (INT; n = 100) or to an active comparison condition (n = 100) consisting of group therapy and case management (GCM). The INT condition will consist of individually administered HIV preventive intervention for adolescent girls involved in the juvenile justice system that integrally addresses delinquency, drug abuse, and trauma exposure, along with group-based training and support for parents. The girl and parent components will run concurrently for three months. The GCM condition will consist of group therapy and case management for girls provided as usual by the juvenile justice department. We will examine intervention effects on proximal outcomes measured at 12 months, the effects of childhood adversity on proximal outcomes, and the mediation of intervention effects. Longer term outcomes will be measured at 24 months. Data will be collected through in-person interviews and questionnaires from focal participants and their parents, official arrest records, and urinary analysis.

ELIGIBILITY:
Inclusion Criteria:

* female, age 13-18 years
* living in Lane County, Oregon
* living at home (biological/adoptive, foster, or other relative care)
* at least one criminal referral and on probation or a formal accountability contract with the juvenile justice system
* documented drug use from juvenile justice risk assessment
* traumatic exposure
* no imminent plans to be placed in out-of-home care

Exclusion Criteria:

* meet criteria for posttraumatic stress disorder

Ages: 13 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 416 (Actual)
Dates: Start 2013-09; Primary Completion 2018-08 (Actual); Study Completion 2020-05 (Actual)

PRIMARY OUTCOMES:
Reduction in HIV/STIs risk behavior in delinquent girls | Baseline and post intervention (6 mos); 12 & 24 month follow-ups
  Girls in the intervention condition are expected to have significantly lower rates of HIV/STI risk behaviors compared to girls in the control condition at each of the time-points post-baseline. Data will be collected through in-person interviews and questionnaires from focal participants and their parents.

SECONDARY OUTCOMES:
Reduction in criminal offending | Baseline and post intervention (6 mos); 12 & 24 month follow-ups
  Girls in the intervention condition are expected to have significantly lower rates of criminal offending behavior compared to girls in the control condition at each of the time points post-baseline. Data will be collected through in-person interviews and questionnaires from focal participants and their parents and official arrest records.

OTHER OUTCOMES:
Reduction in substance use | Baseline and post intervention (6 mos); 12 & 24 month follow-ups
  Girls in the intervention condition are expected to have significantly lower rates of substance use compared to girls in the control condition at each of the time-points post-baseline. Data will be collected through in-person interviews and questionnaires from focal participants and their parents and urinary analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Dana K Smith, PhD, Principal Investigator — Oregon Research Institute
Locations (1):
- Oregon Research Institute, Eugene, Oregon, United States